CLINICAL TRIAL: NCT04266808
Title: Interactive Telehealth and Auto-Biofeedback Sensor System for Individuals Who Use a Wheelchair: Phase II
Brief Title: Interactive Telehealth for Wheelchair Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rancho Research Institute, Inc. (Other)
Collaborators: BioSensics (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sara Mulroy, Research Director, Rancho Research Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R44AG059275-04 (NIH); 5R44AG059275-04 (NIH)
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Spinal Cord Injuries; Paraplegia; Pressure Ulcer, Buttock
Keywords: Spinal cord injury; Pressure Ulcer
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Randomized trial with one intervention arm and one control arm.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessors for both skin integrity and psychosocial measures will be blinded to participants' group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- An interactive telehealth monitoring and biofeedback system (Experimental): Participants in this group will receive feedback of pressure relief maneuvers and wheelchair propulsion activity. Feedback for pressure relief will include information during the activity to identify adequate duration and magnitude of pressure relief activity, reminders of when the next pressure relief is due, and daily aggregate information regarding the number of successful pressure relief maneuvers performed.
  Interventions: Device: An interactive telehealth monitoring and biofeedback system
- Education Control (Sham Comparator): Participants will receive education on the importance and recommended frequency of pressure relief maneuver for prevention of pressure ulcer/injury and on the importance and recommended amounts of physical activity for health.
  Interventions: Behavioral: Education Control

INTERVENTIONS:
Device: An interactive telehealth monitoring and biofeedback system — A pressure sensitive mat located under the user's wheelchair seat cushion and a wheelchair propulsion monitoring device attached to the chair which are interfaced with a phone App based user interface to provide feed back to promote physical activity and pressure relief maneuver performance among wheelchair users.
  Arms: An interactive telehealth monitoring and biofeedback system
Behavioral: Education Control — Participants will receive education on importance of pressure relief maneuvers and physical activity and the recommended amounts of each for prevention of pressure ulcer/injury and for physical health.
  Arms: Education Control

SUMMARY:
During typical daily activity, people with established spinal cord injury perform significantly fewer pressure-relief maneuvers than the recommended frequency while overestimating their adherence on recall surveys of pressure relief activity. The rate of pressure ulcer recurrence in individuals with a prior ulcer is 44% in those with surgical repair and as high as 75% in those with non-surgical healing indicating that increased attention to pressure relief is critical for these individuals.This study will evaluate the efficacy of a wheelchair sensor and app-based biofeedback for establishing healthy self-management behaviors (pressure relief maneuvers and daily physical activity). Investigators will enroll 50 participants with paraplegia from spinal cord injury who use a manual wheelchair for mobility and have a history of pressure ulcer that has healed or is six months post-surgical repair. Participants will be randomized into one of two groups: an intervention group that will receive an education intervention and the proposed technology to be used for one year, and a control group that will receive only the education intervention. The primary outcome will be pressure ulcer occurrence over one year. Investigators hypothesize that participants receiving the intervention of biofeedback on their pressure relief activity will have a lower recurrence of pressure ulcer than the education only control group. Secondary outcomes include depressive symptoms, self-efficacy, participation and satisfaction with life. Investigators hypothesize that increasing physical activity will reduce depressive symptoms and improve participation and satisfaction with life.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to evaluate the efficacy of an interactive tele-health monitoring and biofeedback system to establish healthy behaviors and promote self-management of pressure relief maneuvers and physical activity.

Procedures and Course of Study:

Baseline 50 participants will be enrolled. At study entry participants will complete four baseline questionnaires and have a Nurse Practitioner or Physician's Assistant inspect their ischial skin to ensure that their prior ulcer is fully healed. A pressure-sensing mat (PRESS) will be placed under their wheelchair cushion, and a wheelchair propulsion motion sensor (WAMS) will be placed on the rear wheel of their wheelchair. The PRESS and WAMS sensors will record participants' pressure relief and wheelchair propulsion activity for the next two weeks.

Intervention:

Participants will then return to the clinic and the study physical therapist will provide all participants with education on importance of pressure relief maneuvers and physical activity for health as well as training in the 3 styles of pressure relief (forward and side leans, depression raise) and shoulder strengthening exercises to protect against shoulder impingement and pain with increased pressure relief and wheelchair propulsion activity. The study physical therapist will then assist all participants in setting goals to increase pressure relief frequency and/or duration and wheelchair propulsion pushes for the future based on their baseline activity. Participants will be randomized into one of two groups: feedback and no feedback. In both groups pressure relief and wheelchair propulsion activity will be recorded by the PRESS and WAMS sensors for the 12 months. Those participants in the no-feedback group will have the feedback features of the system disabled. Those participants in the feedback group will receive instant visual feedback on pressure relief duration and daily summary charts for both pressure relief and wheelchair propulsion activities.

Follow-up:

Every month following the intervention for 12 months, a physical therapist will contact participants by phone to inquire whether their ischial skin integrity has changed and whether they have developed a pressure ulcer. Additionally, all participants will return to the clinic at 3, 6, 9, and 12 months after the intervention and a nurse practitioner will examine their ischial skin and review their medical records to determine if a pressure ulcer has developed. Participants will repeat the 4 questionnaires from the baseline evaluation at each follow-up visit. At the 12 month follow-up visit, participants will return the sensor equipment.

ELIGIBILITY:
Inclusion Criteria:

* paraplegia from Spinal Cord Injury
* a history of pressure ulcer that has healed or 6 months post surgical repair
* use a manual wheelchair for mobility
* able to perform pressure relief maneuvers independently

Exclusion Criteria:

* unable/unwilling to return to clinic for follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Pressure Ulcer | Any time during the one year active phase of the study intervention
  Any stage of Pressure Ulcer/Injury identified in the ischial region
Change in mean number of cycles of self-propulsion per day from Baseline | The four weeks preceding the 12 month assessments
  The increase or decrease in number of cycles of self-propulsion per day over the 4 weeks preceding the 12 month assessment
Change in mean number of pressure relief maneuvers per day from Baseline | The four weeks preceding the 12 month assessments
  The increase or decrease in mean number of pressure relief maneuvers per day over the 4 weeks preceding the 12 month assessment from Baseline
Time to Recurrence of Pressure Ulcer | Any time during the one year active phase of the study intervention
  The number of days from study entry to identification of recurrence of Pressure Ulcer/Injury

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 score | 12 months
  Change in Questionnaire scores measuring depressive symptoms at 12 month assessment from baseline score
Change in University of Washington Self Efficacy Short Form | 12 months
  Change in scores on Questionnaire measuring self-efficacy at 12 month assessment from baseline score
Change in Reintegration to Normal Living Index | 12 months
  Change score on Questionnaire measuring participation at 12 month assessment from baseline score
Change in Satisfaction with Life Scale | 12 months
  Change in score on Questionnaire measuring satisfaction with life at 12 month assessment from baseline score

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mulroy, PhD, PT, Principal Investigator — Rancho Los Amigos National Rehab Ce
Locations (1):
- Rancho Los Amigos National Rehabilitaiton Center, Downey, California, United States

IPD SHARING:
Plan to Share IPD: No